CLINICAL TRIAL: NCT06166563
Title: Effects of Indoor Activity on the Integrity and Function of the Intestinal Barrier of Patients With Fibromyalgia and Irritable Bowel Syndrome
Brief Title: Exercise, Irritable Bowel Syndrome and Fibromyalgia
Acronym: AF-IBS-FM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Francesco Russo, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF-FM 01
Record Dates: First submitted 2023-11-24; First posted 2023-12-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome
Keywords: Fibromyalgia; Irritable Bowel Syndrome; Exercise; Gastrointestinal Functions; Physical Activity
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AF-FM (Active Comparator): Patients with Fibromyalgia
  Interventions: Behavioral: Exercise Program
- AF-IBS (Active Comparator): Patients with irritable bowel syndrome
  Interventions: Behavioral: Exercise Program
- AF-FM-IBS (Active Comparator): Patients with fibromyalgia and irritable bowel syndrome
  Interventions: Behavioral: Exercise Program

INTERVENTIONS:
Behavioral: Exercise Program — The intervention includes an individualized exercise program in Frequency, Intensity, Time, and Type (FITT).

SUMMARY:
The project focuses on "somatic functional syndrome", a category of disorders characterized by subjective symptoms, suffering and disability without evident organic or functional alterations. Syndromes such as Fibromyalgia, Irritable Bowel, Chronic Fatigue and Restless Legs fall into this category. Patients seek diagnoses and treatments, often consulting multiple doctors. The proposed alternative approach involves physical activity as the cornerstone of therapy, with a focus on fibromyalgia.

Fibromyalgia manifests itself with musculoskeletal pain, chronic fatigue, sleep disturbances and other symptoms. The text highlights a correlation between fibromyalgia and gastrointestinal disorders, in particular Irritable Bowel. Both syndromes share pathophysiological mechanisms, including alteration of intestinal permeability and psychosocial factors.

An important note is the possible compromise of the integrity of the intestinal wall, with consequences on general health. Inflammation, dysbiosis, and altered intestinal permeability contribute to a vicious cycle that can lead to cardiovascular, neurodegenerative, and inflammatory diseases.

Regular physical activity is a possible improvement for fibromyalgia symptoms, with scientific studies demonstrating its effectiveness. A sedentary lifestyle is linked to gastrointestinal problems, and physical exercise can promote gastrointestinal motility and counteract disorders such as gastric reflux and irritable bowel syndrome.

The research aims to focus on the effects of physical activity on gastrointestinal and extra-gastrointestinal symptoms in patients with fibromyalgia and irritable bowel disease. The effects on intestinal integrity, dysbiosis and markers of inflammation are also examined. The research also aims to evaluate the psychological aspects of these syndromes.

DETAILED DESCRIPTION:
Patient Recruitment: the study protocol has been designed as a prospective, single-center, active-agent-controlled comparison in parallel groups of adult outpatients (18-65 years) affected by:

1. fibromyalgia (FM), from the "Rheumatology" Clinic of the National Institute of Gastroenterology "S de Bellis" Castellana G;
2. irritable bowel syndrome (IBS), from the "Celiac Disease and Functional Disorders" Clinic of the National Institute of Gastroenterology "S de Bellis" Castellana G;
3. both comorbidities (FM+IBS) from the above-cited clinics. The patients will also be recruited among the fibromyalgia patients registered with the "Smile Association" of Castellana G. (BA).

Information regarding the participant's health status will be gathered through a comprehensive visit, encompassing an interview covering lifestyle, medical history, and a physical examination. Additionally, metabolic parameters, including blood sugar, HbA1c, lipid profile, and body weight, must fall within the normal range of values. Before providing written consent, all participants will receive verbal and written details of the study. The recruitment and evaluation of patients will be structured into the following phases:

V1. (Day -14): Patients will be briefed on the study and consent to it. A clinical anamnestic form will be filled out to account for the influence of current medications. For the next 14 days, participants will keep a daily symptom diary, noting stool characteristics with the Bristol scale and evaluating intestinal habits.

V2. (Day 0): Patients will return for blood sampling and the collection of essential biological samples (urine, feces) required for laboratory evaluations as specified by the study. Additionally, they will fill out questionnaires on gastrointestinal (GI) and fibromyalgia (FM) symptoms. During this visit, psychological, quality of life (QoL), physical activity assessments and anthropometric and bioimpedance measurements will be conducted. Field tests to gauge physical fitness will be performed. Patients will receive instructions, supported by specialized personnel, to follow a specific indoor physical activity regimen. Every four weeks, the same field tests from V2 will be conducted to monitor the effectiveness of the work protocol.

V3. (Day 120): Patients will again complete questionnaires on GI symptoms, FM symptoms, psychological symptoms, QoL, and physical activity level. Physical activity (PA) parameters will be collected, and any adverse events during the intervention will be evaluated. Finally, blood and biological samples necessary for the laboratory evaluations required by the study will be taken.

Evaluation of FM Symptoms: The assessment of FM symptoms involves utilizing a series of validated questionnaires, some specific to FM and others more general (i.e., Fibromyalgia Impact Questionnaire, modified version (FIQ-R); Digital Tender Point examination).

Evaluation of GI Symptoms: A patient's clinical history form is completed before assessing GI symptoms. Subsequently, two questionnaires are administered: the IBS-SSS, specific to IBS symptoms.

Psychological Assessment: The psychological profile is assessed using validated questionnaires. Initially, a history form identifies prior psychopathological disorders or family history. Additionally, first and second-level stress factors linked to symptoms are pinpointed. At baseline and day 120, participants complete pre- and post-administered psychological questionnaires covering various aspects, including the Symptom Checklist (SCL)-90-R, Perceived Stress Scale (PSS), World Health Organization Quality of Life-Brief (WHOQOL-Brief), Delaying Gratification Inventory (DGI), Rotter's Locus of Control Scale, Subjective Happiness Scale (SHS), Attachment Style Questionnaire (ASQ), and Psychological Well-Being Scales (PWBS).

Anthropometric and Bioimpedance Assessment: The subjects' physical characteristics (body weight, height, circumferences) are assessed through direct measurement. Bioimpedance measurement involves a non-invasive, rapid, and quickly executed examination, ideal for measuring nutritional status (lean mass, fat mass, cellular and muscle mass), hydration status (water retention, swelling, hyperhydration, inflammation), basal metabolism, and "ideal weight".

Evaluation of Intestinal Permeability (IP): IP will be evaluated at baseline (day 0) and day 120. This involves administering a mixture of 40 g sucrose, 10 g lactulose, 5 g mannitol, and 1 g sucralose and measuring their gastrointestinal (GI) absorption through urinary excretion of these sugars. Urine will be collected over the next 5 hours in containers with added chlorhexidine (500 µL) as a preservative. The different sugars in the urine will be determined using high-pressure liquid chromatography (HPLC) and subsequent pulsed amperometric detection. Results will be expressed as a percentage of the excreted sugars in urine relative to the administered amount.

Barrier Peptide Assay: Zonulin, intestinal fatty acid binding protein (I-FABP), diamine oxidase (DAO), and D-lactate assays will be conducted at baseline (day 0) and day 120 using commercially available Enzyme-Linked Immunosorbent Assay (ELISA) methods.

Intestinal Microbiota Analysis: The evaluation of the intestinal microbiota involves extracting total bacterial metagenomic DNA from fecal samples. Microbiome characterization will be performed using a DNA metabarcoding approach and shotgun metatranscriptomic. DNA metabarcoding analysis will use the V5-V6 hypervariable regions of the 16S rRNA for bacteria (MiSeq-Illumina platform). Significant samples in the DNA metabarcoding analysis will undergo metatranscriptomic analysis (NextSeq 500 platform - Illumina). Metagenomic and metatranscriptomic data will be analyzed using bioinformatics pipelines.

Indole and Skatole Assay: Indole will be assayed using a colorimetric analytical method, while skatole will be assessed using a refined chromatographic method with fluorimetric detection. Both assays will be conducted on a urine sample. This investigation will be conducted at baseline and day 120.

Biochemical analyses: blood levels of interleukin (IL)-6, IL-8, IL-10, tumor necrosis factor (TNF)-alpha, and peptides involved in the regulation of GI motility (somatostatin, motilin, serotonin, somatostatin, motilin, serotonin, etc.) will be assayed in blood samples at baseline (day 0) and day 120 using ELISA methods.

Physical Activity Assessment: To assess the level of physical activity, the International Physical Activity Questionnaire (IPAQ short-form) will be administered before initiating the intervention protocol. Additionally, participants will be asked to wear an accelerometer [V1], provided to them on the day of enrollment and modeled for the subsequent seven days.

Before starting the intervention protocol at the end of each month (4 weeks), field tests will be conducted to assess the physical fitness status of the subjects: a) Two-Walking test/ 6-min Walking test; b) Hand Gripp Test; c) Sit and Reach Test.

However, special precautions must be considered when conducting field tests for individuals with FM. Namely, A) symptoms before the test will be examined to determine the severity and location of pain and the individual's level of fatigue. B) The individual's previous and current exercise experience will be assessed to determine the likelihood of increased symptoms after the test. C) High levels of motivation using constant verbal encouragement for the individual to reach their maximum level will be provided during the test D) Adequate rest and recovery for different physiological systems and muscle groups will be allowed between tests. E) Pain and fatigue levels will be continuously monitored during tests. F) Before tests and workouts, individuals will be informed about the differences between soreness and fatigue after exercise and the normal fluctuations of pain and fatigue due to FM. G) The test will be chosen based on the subject's conditions (as recommended by the American College of Sports Medicine). The same operator will repeat the most suitable test under the same conditions at the end of each cycle. Typically, the 6-minute Walking test is most convenient for these subjects. For subjects with IBS, the intervention protocol remains the same, but the parameter of aerobic activity intensity will be adjusted, starting from 40-60% of HR up to a maximum of 75%.

Treatment Physical Activity: Individuals with FM exhibit reduced aerobic capacity and muscle function (i.e., strength and endurance), diminished functional performance (e.g., walking, climbing stairs) and physical fitness. These reductions are generally attributed to widespread chronic pain that limits the individual's ability to complete daily activities. However, regular, low-impact physical exercise is valuable in breaking the cycle of chronic pain, increasing fatigue resistance, acting on psychophysical stress, and improving QoL. Physical exercise enhances Flexibility, Neuromuscular function, Cardiorespiratory function, Functional performance, Blood pressure levels (BP), Pain and other FM symptoms, Self-efficacy, Depression, and Anxiety. Due to potential pain and symptom exacerbation, the subject's medical history and health status must be examined before conducting field tests or prescribing an exercise program. Objective assessment of physiological and functional limitations will allow for optimal testing and training.

Intervention Protocol:

Frequency: Combined physical exercise (aerobic, resistance, and flexibility activities) will be performed inside a gym whose characteristics are detailed at the end of the document (see "Indoor Physical Activity Gym Characteristics") twice a week for the first weeks, gradually increasing to three times a week, on non-consecutive days, for 120 days.

Intensity: Physical activity intensity will be monitored using a heart rate monitor and personalized through the Tanaka formula. The "TALK TEST" will also measure pace, and the BORG scale will measure fatigue perception.

Initially, the intensity of the aerobic activity will be low (30% heart rate - HR - max) and progressively increase to moderate intensity (40-60% HR max); for resistance/strength exercises, the intensity will range from 40-80% 1- Repetition Maximum (RM) to 60-80% 1-RM. Flexibility exercises will always consider the Range of Motion (ROM) and be limited to pain-free movements.

Type: The type of physical activity is moderate aerobic with the addition of resistance and flexibility exercises.

Aerobic activity: low-impact/exercise without load to minimize potential exercise-induced pain.

Resistance activities: exercises with elastic bands, dumbbells, wrist or ankle weights, exercises with isotonic machines, or bodyweight exercises.

Flexibility exercises: stretching exercises with elastic bands and without load.

A single 60-minute session will be structured as follows: Warm-up, Walking (aerobic activity); Strength/resistance exercises, Flexibility exercises; and Cool-down.

Time: Aerobic activity: initially 10 minutes, gradually increasing to 30-60 minutes per session.

Strength exercises: progressive increase from 4-5 to 8-12 repetitions, moving from 2 to 4 sets per muscle group with a 2-3 minutes' rest between sets.

Flexibility exercises: maintaining the stretch, initially for 10-30 seconds, up to over 60 seconds.

Exercise volume will be reduced if symptoms increase during or after exercise. Reducing intensity or duration before lowering frequency may help maintain a regular PA pattern. All activities will be supervised by Doctors in Sciences and Techniques of Preventive and Adaptive Motor Activities.

Primary Endpoint: Perceived physical function will be evaluated using the total FIQ-R score (higher scores indicate worse functioning). The expected result is a 20% improvement in the total FIQ-R score at the end of the intervention.

Secondary Endpoints: The relationship between FIQ-R and IBS-SSS, which investigates the severity of GI symptoms about PI, will be evaluated. The effects of indoor physical activity on psychological, nutritional, inflammatory, and dysbiosis profiles will also be investigated.

Statistical Analysis: Data will be presented as mean (SD) or median and 5th and 95th percentiles, depending on whether they are continuous or categorical variables. All comparisons will be made using non-parametric tests to avoid assumptions of normal data distribution. Proportions related to dichotomous variables will be compared using the X2 test. Values of P <0.05 at two tails will be considered statistically significant. All patients receiving physical activity instructions will be included in the statistical analysis for data comparison at the end of the treatment period, and dropouts will be categorized as non-responders (Intention to Treat analysis). The comparison between data at the end of the intervention period and the baseline will be performed, considering only those who have completed the intervention (per protocol analysis). All statistical analyses will be performed using the SigmaSTAT statistical package (Systat Software, Inc., San Jose, California, USA) and the GraphPad Prism 5 package (GraphPad Software Inc., La Jolla, California, USA). Questionnaire data will be entered into a database by someone not involved in the study.

Study Power Calculation: The sample size is calculated to detect a 20% improvement in the total FIQ-R score before and after the intervention. Considering a standard deviation of 30, a power of 0.80, and a significance level of 0.05, a minimum of 44 patients per group must be recruited. With a 25% dropout, each group will comprise 55 patients (a total number of 165).

ELIGIBILITY:
Inclusion Criteria:

* Satisfaction of the ACR diagnostic criteria for the diagnosis of FM,
* A total Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) score of ≥ 125 (moderate to severe IBS symptoms) for the satisfaction of the Rome III-IV criteria in patients with IBS.

Exclusion Criteria:

* Serious cardiac, hepatic, neurological, psychiatric, or gastrointestinal diseases other than IBS (e.g., inflammatory bowel disease, diverticular disease/diverticulitis) that could explain the current symptoms.
* Specific therapy for symptoms due to pathologies (educational programs, alternative medicine, psychotherapy). In the case of subjects who were previously undergoing treatment, they may participate in the study provided they suspend the ongoing therapy until the symptoms reappear.
* The use of drugs to treat FM and IBS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
IBS symptoms assessment | At baseline and day 120
  To evaluate the effectiveness of an exercise intervention on IBS symptoms as measured by a change in the IBS-Symptom Severity Scale (IBS-SSS) questionnaire score from baseline.
  The IBS-SSS is a validated questionnaire for gastrointestinal symptoms and provides a global measure of symptom severity by assessing five items ("severity of abdominal pain", "frequency of abdominal pain", "severity of abdominal distension", "dissatisfaction with bowel habits", "impact of symptoms on quality of life") on a visual analog scale. The values of the five items are added together to give a total score between 0 and 500. Cases are then classified as 'mild' (75 to 175), 'moderate' (175 to 300) and 'severe' (>300).
Fibromyalgia symptom assesment | At baseline and day 120
  To evaluate the effectiveness of an exercise intervention on IBS symptoms as measured by a change in the Fibromyalgia Impact Questionnaire, modified version (FIQ-R) scores from baseline.
  The FIQ serves as a tool for assessing and evaluating the condition of patients with fibromyalgia (FM) and tracking their progress and outcomes. Specifically designed to gauge the aspects of health status most impacted by FM, the FIQ comprises ten items. The initial item consists of 11 questions about physical functioning, each rated on a 4-point Likert-type scale. The subsequent items (2 and 3) prompt patients to indicate the number of days they felt well and the days they were unable to engage in work or housework due to FM symptoms. Items 4 through 10 feature horizontal linear scales with ten increments, allowing patients to rate work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression.

SECONDARY OUTCOMES:
Psychological Assessment: | At baseline and day 120
  The Symptom Checklist (SCL)-90-R questionnaire will evaluate the psychological profile
  The Symptom Checklist-90-Revised (SCL-90-R) is a widely employed self-report questionnaire in clinical and research settings. It aims to evaluate diverse psychological symptoms and distress in individuals. Comprising 90 items, the SCL-90-R addresses dimensions of psychological well-being and psychopathology, including somatization, obsessive-compulsive symptoms, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. Respondents use a Likert scale ranging from 0 (not at all) to 4 (extremely) to rate the extent of their experience with each symptom over a specified timeframe, typically the past week. This questionnaire offers a comprehensive profile of an individual's psychological symptoms, aiding in identifying areas of distress or dysfunction.
Gastroduodenal permeability | At baseline and day 120
  Gastroduodenal permeability will be assessed by administering a mixture of sucrose-lactulose-mannitol-sucralose and measuring their gastrointestinal absorption by urinary excretion of these sugars
Evaluation of Barrier Peptide Integrity | At baseline and day 120
  Zonulin, I-FABP, DAO, and D-lactate assays will be performed using commercially available ELISA assays for each peptide.
Intestinal microbiota analysis | At baseline and day 120
  Any differences in the intestinal microbial population in the different disease patterns considered will be evaluated using appropriate genetic and molecular investigations (Illumina/Solexa Genetic Analyzer HiSeq) on the patient's stool samples.
Evaluation of Intestinal dysbiosis | At baseline and day 120
  The intestinal dysbiosis will be evaluated by assaying Indole using a colorimetric analytical method as a marker of fermentative dysbiosis, Skatole, a marker of putrefactive dysbiosis, will be assessed using a refined chromatographic method with fluorimetric detection. Both assays will be conducted on a urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Russo, Principal Investigator — National Institute for Digestive Diseases IRCCS " Saverio de Bellis"
Locations (1):
- IRCCS Saverio de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster C, Porcari JP, Anderson J, Paulson M, Smaczny D, Webber H, Doberstein ST, Udermann B. The talk test as a marker of exercise training intensity. J Cardiopulm Rehabil Prev. 2008 Jan-Feb;28(1):24-30; quiz 31-2. doi: 10.1097/01.HCR.0000311504.41775.78. PMID 18277826
- [Background] Jones KD, Clark SR, Bennett RM. Prescribing exercise for people with fibromyalgia. AACN Clin Issues. 2002 May;13(2):277-93. doi: 10.1097/00044067-200205000-00012. PMID 12011599
- [Background] Kingsley JD, McMillan V, Figueroa A. The effects of 12 weeks of resistance exercise training on disease severity and autonomic modulation at rest and after acute leg resistance exercise in women with fibromyalgia. Arch Phys Med Rehabil. 2010 Oct;91(10):1551-7. doi: 10.1016/j.apmr.2010.07.003. PMID 20875513
- [Background] Mannerkorpi K, Iversen MD. Physical exercise in fibromyalgia and related syndromes. Best Pract Res Clin Rheumatol. 2003 Aug;17(4):629-47. doi: 10.1016/s1521-6942(03)00038-x. PMID 12849716
- [Background] Rooks DS. Talking to patients with fibromyalgia about physical activity and exercise. Curr Opin Rheumatol. 2008 Mar;20(2):208-12. doi: 10.1097/BOR.0b013e3282f5687a. PMID 18349753
- [Background] Tanaka H, Monahan KD, Seals DR. Age-predicted maximal heart rate revisited. J Am Coll Cardiol. 2001 Jan;37(1):153-6. doi: 10.1016/s0735-1097(00)01054-8. PMID 11153730
- [Background] Valkeinen H, Alen M, Hannonen P, Hakkinen A, Airaksinen O, Hakkinen K. Changes in knee extension and flexion force, EMG and functional capacity during strength training in older females with fibromyalgia and healthy controls. Rheumatology (Oxford). 2004 Feb;43(2):225-8. doi: 10.1093/rheumatology/keh027. Epub 2003 Sep 16. PMID 13130154
- [Background] Valkeinen H, Hakkinen A, Hannonen P, Hakkinen K, Alen M. Acute heavy-resistance exercise-induced pain and neuromuscular fatigue in elderly women with fibromyalgia and in healthy controls: effects of strength training. Arthritis Rheum. 2006 Apr;54(4):1334-9. doi: 10.1002/art.21751. PMID 16575859
- [Background] Wilson RC, Jones PW. A comparison of the visual analogue scale and modified Borg scale for the measurement of dyspnoea during exercise. Clin Sci (Lond). 1989 Mar;76(3):277-82. doi: 10.1042/cs0760277. PMID 2924519
- [Background] Linsalata M, Riezzo G, D'Attoma B, Clemente C, Orlando A, Russo F. Noninvasive biomarkers of gut barrier function identify two subtypes of patients suffering from diarrhoea predominant-IBS: a case-control study. BMC Gastroenterol. 2018 Nov 6;18(1):167. doi: 10.1186/s12876-018-0888-6. PMID 30400824
- [Background] Barsky AJ, Borus JF. Functional somatic syndromes. Ann Intern Med. 1999 Jun 1;130(11):910-21. doi: 10.7326/0003-4819-130-11-199906010-00016. PMID 10375340
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Martinez-Lavin M. Biology and therapy of fibromyalgia. Stress, the stress response system, and fibromyalgia. Arthritis Res Ther. 2007;9(4):216. doi: 10.1186/ar2146. PMID 17626613
- [Background] Akkaya N, Akkaya S, Atalay NS, Balci CS, Sahin F. Relationship between the body image and level of pain, functional status, severity of depression, and quality of life in patients with fibromyalgia syndrome. Clin Rheumatol. 2012 Jun;31(6):983-8. doi: 10.1007/s10067-012-1965-9. Epub 2012 Mar 7. PMID 22395855
- [Background] Sarzi-Puttini P, Giorgi V, Marotto D, Atzeni F. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. Nat Rev Rheumatol. 2020 Nov;16(11):645-660. doi: 10.1038/s41584-020-00506-w. Epub 2020 Oct 6. PMID 33024295
- [Background] Kim YS. Why should gastroenterologists know about fibromyalgia? Common pathogenesis and clinical implications. J Neurogastroenterol Motil. 2011 Jan;17(1):1-3. doi: 10.5056/jnm.2011.17.1.1. Epub 2011 Jan 26. No abstract available. PMID 21369484
- [Background] Johannesson E, Jakobsson Ung E, Sadik R, Ringstrom G. Experiences of the effects of physical activity in persons with irritable bowel syndrome (IBS): a qualitative content analysis. Scand J Gastroenterol. 2018 Oct-Nov;53(10-11):1194-1200. doi: 10.1080/00365521.2018.1519596. Epub 2018 Nov 25. PMID 30472905
- [Background] Russo F, Riezzo G, Linsalata M, Orlando A, Tutino V, Prospero L, D'Attoma B, Giannelli G. Managing Symptom Profile of IBS-D Patients With Tritordeum-Based Foods: Results From a Pilot Study. Front Nutr. 2022 Feb 15;9:797192. doi: 10.3389/fnut.2022.797192. eCollection 2022. PMID 35242794
- [Background] Russo F, Riezzo G, Orlando A, Linsalata M, D'Attoma B, Prospero L, Ignazzi A, Giannelli G. A Comparison of the Low-FODMAPs Diet and a Tritordeum-Based Diet on the Gastrointestinal Symptom Profile of Patients Suffering from Irritable Bowel Syndrome-Diarrhea Variant (IBS-D): A Randomized Controlled Trial. Nutrients. 2022 Apr 8;14(8):1544. doi: 10.3390/nu14081544. PMID 35458106